CLINICAL TRIAL: NCT05382052
Title: Study of ctDNA as Prognostic Factor on Resectable Stage IIIA NSCLC Patients Treated With Neoadjuvant Treatment
Acronym: REAL-NADIM
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 21/05_REAL-NADIM
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer Stage III; Neoadjuvant Treatment
Keywords: Resectable stage IIIA; ctDNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Five blood samples per patient will be collected:
  * Before starting neoadjuvant treatment
  * At the end of the neoadjuvant treatment and before the surgery
  * After surgery
  * 6 months after surgery
  * At first disease progression (if occurs within 24 months after surgery)
  The blood samples (5-10 ml each) will be collected in two Cell-Free DNA BCT tube and two PTT EDTA K2.
  These samples will be sent to the central laboratory the same day of extraction at room temperature.
  ctDNA will be extracted using the QIAamp Circulating Nucleic Acid Kit. NGS analysis of ctDNA will be performed using a panel that will target at least of 1.5 Mb and will include genes of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The study is based on a blood sample analysis in stage IIIA non-small lung cancer patients that are going to receive neoadjuvant treatment in the real world. The patients participating in this non-interventional study will not receive treatment in relation to the study. Prospective information about treatment after neoadjuvant treatment and after the last blood extraction will not be collected.

SUMMARY:
This is an observational, prospective, multicentre and nationwide study.

The study enroll resectable stage IIIA non-small cell lung cancer patients that are going to receive neoadjuvant treatment in real world.

The primary objective of this study is evaluating whether there is a significant association between ctDNA clearance (no detection of ctDNA) after neoadjuvant treatment and before surgery and progression free survival.

DETAILED DESCRIPTION:
This is an observational, multicenter, one-arm, non-comparative, prospective study that will not under any circumstances interfere in the physician's normal clinical practice. Being limited to the collection of blood samples at five times and patient data, it does not entail any diagnostic or therapeutic procedure outside of normal clinical practice.

Approximately 100 resectable stage IIIA non-small cell lung cancer patients that are going to receive neoadjuvant treatment in real world will be recruited for this study in Spain. With this figure, it can be estimated whether ctDNA, both baseline and its negativization, has a role as a prognostic marker in the evolution of these patients in real-life conditions.

The primary objective of this study is evaluate whether there is a significant association between ctDNA clearance (no detection of ctDNA) after neoadjuvant treatment and before surgery and progression free survival.

The study is planned with the recruitment of patients over a year to a follow-up of 36 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Previously untreated patients with histologically- or cytologically- documented NSCLC who present stage IIIA disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology) and also, potentially resectable locally advanced NSCLC patients' stage IIIB with T3N2 disease according to 8th edition can be included.
* 2. Tumor should be considered resectable before study entry by a multidisciplinary team
* 3. ECOG 0-1
* 4. Age ≥ 18 years at time of study entry
* 5. Patients that are going to be treated with neoadjuvant treatment before surgery
* 6. Patient capable of proper therapeutic compliance and accessible for correct follow-up
* 7. Patients must have signed, dated and IRB/EC-approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.

Exclusion Criteria:

* 1. Patients who refuse to sign and date an IRB/IEC-approved written informed consent form.
* 2. No possibility of venipuncture
* 3. Any medical, mental, or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable stage IIIA non-small cell lung cancer patients that are going to receive neoadjuvant treatment in real world.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether there is a significant association between ctDNA clearance after neoadjuvant treatment and before surgery and progression free survival (PFS). | From date of end of neoadjuvant treatment and before surgery until the date of progression free survival, assessed up to 24 months
  To assess the association between the baseline ctDNA and ctDNA clearance with each one of the three outcomes: after neoadjuvant treatment, before surgery and PFS

SECONDARY OUTCOMES:
To evaluate whether there is a significant association between ctDNA clearance after neoadjuvant treatment and before surgery and overall survival. | From date of end of neoadjuvant treatment and before surgery until the date of death, assessed up to 24 months
  To assess the association between the baseline ctDNA and ctDNA clearance with each one of the three outcomes: after neoadjuvant treatment, before surgery and Overall Survival
To evaluate whether there is a significant association between ctDNA clearance and pathological complete response or major pathologic response. | From the end of neoadjuvant treatment and before surgery until the death of complete response or MPR, assessed up to 24 months
  To assess the association between the baseline ctDNA and ctDNA clearance with each one of the two outcomes: after complete response or major pathologic response (MPR).
To identify somatic mutations in ctDNA that predispose to a better/worse overall survival | From the date of extraction of blood in pretreatment period until the date of major pathologic response or death, assessed up to 24 months
  To identify somatic mutations in ctDNA in the pre-treatment plasma that predispose to a better/worse overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — President of Grupo Español de Cáncer de Pulmón
Locations (20):
- Spain (20):
  - Hospital Universitario De A Coruna, A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital De Basurto, Bilbao, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - ICO Girona, Hospital Josep Trueta, Girona, Girona
  - Complejo Hospitalario de Navarra, Pamplona, Iruña
  - Hospital Universitario de Jaén, Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario la Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Regional de Málaga, Málaga, Málaga
  - Hospital Universitari Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Web page of the sponsor where users can find more information about Fundacion GECP studies. — http://www.gecp.org